CLINICAL TRIAL: NCT02201810
Title: Enhancing the Efficacy of Smoking Quit Line in the Military
Brief Title: Enhancing the Efficacy of Smoking Quit Line in the Military (AFIII Renewal)
Acronym: Freedom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: University of Tennessee (Other)
Responsible Party: Principal Investigator, Melissa Little, PhD, MPH, Associate Professor, Department of Public Health Sciences, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FWH20140076H
Record Dates: First submitted 2014-07-24; First posted 2014-07-28 (Estimated); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Initial Efficacy of Quit Line; Efficacy of Secondary Reengagement Intervention
Keywords: smoking cessation; quit line; nicotine replacement therapy; tobacco intervention
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 2nd level intervention: Rate Reduction (Experimental): Rate reduction intervention
  Interventions: Behavioral: Rate reduction intervention; Behavioral: Proactive QL
- 2nd level intervention: Recycling (Experimental): Recycling Group
  Interventions: Behavioral: Recycling Group; Behavioral: Proactive QL
- 2nd level intervention: Choice (Experimental): Choice Group
  Interventions: Behavioral: Choice Group; Behavioral: Proactive QL

INTERVENTIONS:
Behavioral: Rate reduction intervention
  Arms: 2nd level intervention: Rate Reduction
Behavioral: Recycling Group
  Arms: 2nd level intervention: Recycling
Behavioral: Choice Group
  Arms: 2nd level intervention: Choice
Behavioral: Proactive QL

SUMMARY:
This study is a randomized clinical trial designed to measure the effectiveness of three QL interventions for smokers who failed to quit an initial smoking cessation intervention, but remain motivated to quit smoking.

DETAILED DESCRIPTION:
In the investigators' previous QL protocol, FWH20080093H, the investigators documented that a military-tailored QL was associated with high rates of sustained smoking cessation. The proactive QL produced superior cessation rates at a one year follow-up compared to a reactive QL. Unfortunately, even with high rates of cessation, a large number of participants (the majority of participants) fail to remain quit at follow-up. Civilian QLs have observed the same marked decay of sustained cessation rates from the end of treatment to the one year follow-up.

An opportunity exists to reengage these smokers who relapse or fail to quit by the end of QL treatment. Civilian QLs use one of two treatments, Recycling (repeat the smoking cessation counseling) or Rate Reduction (cut down over time), as the primary methods for treatment reengagement. Unfortunately, these methods of reengaging the relapsed/failed to quit smoker have not been systematically evaluated. As such, we propose to randomize participants who relapse or fail to quit by the end of the intervention to either (1) repeating the proactive QL (Recycle); (2) smoking reduction with the goal of eventual cessation (Rate Reduction); or (3) the choice of Recycle or Rate Reduction (Choice). Efficacy will be established by assessing both point prevalence and continuous abstinence at a 12 month follow-up.

All participants (approximately 1900) are consented to follow-up treatment reengagement since we do not know a priori who will quit and who will not quit/relapse. The investigators anticipate, based on the investigators' QL study that about 30% will quit and remain quit based on the eight-week proactive QL and about 70% will either not quit or relapse (n≈1300). Those that are smoking at the three-month follow-up are stratified (based on whether they quit and relapsed vs. not quitting at all in the Proactive QL based upon self-report) and randomized to the three treatment reengagement strategies (Recycle, Rate Reduction, or Choice), each one lasting 8 weeks. Then, at one year follow-up, the investigators will assess both point prevalence and continuous abstinence. Since we are intervening on those that initially failed to quit or relapsed, continuous abstinence will be defined from the point of the last treatment reengagement intervention (one year from that point).

ELIGIBILITY:
Inclusion Criteria: To be included, individuals will be

* Active Duty, Retired, or Dependent with Tricare benefits
* Participants must be at least 18 years old
* Smoked five or more cigarettes a day for at least one year
* Live in the 48 contiguous states, Alaska or Hawaii
* Participants must have the ability to understand consent procedures, and have access to a telephone for participation
* Seriously thinking of quitting smoking cigarettes in the next 30 days

Exclusion Criteria:

* Persons who have a known or unknown knowledge of an allergy or hypersensitivity to Nicotine Replacement Therapy (NRT)
* Women who are pregnant, breastfeeding or planning to become pregnant during the next 12 months
* Persons diagnosed with an unstable heart condition will be excluded as NRT is contraindicated in these groups

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 614 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Effectiveness of randomized reengagement interventions | From 3 months follow up to 1 year follow up
  We will assess tobacco status (both 7-day point prevalence and continuous abstinence) at the follow-up period (one year after reengagement interventions are completed) to assess outcome.

SECONDARY OUTCOMES:
One-year outcome from the initially successful group that quit smoking | 1-yr after initial randomization

CONTACTS AND LOCATIONS:
Overall Officials: Robert Klesges, PhD, Principal Investigator — UTHSC; Wayne Talcott, PhD, Principal Investigator — UTHSC
Locations (1):
- Wilford Hall Ambulatory Surgical Center, Lackland Air Force Base, Texas, United States

REFERENCES:
- [Background] Little MA, Ebbert JO, Bursac Z, Talcott GW, Talley L, LeRoy KM, Womack CR, Hryshko-Mullen AS, Klesges RC. Enhancing the efficacy of a smoking quit line in the military: Study rationale, design and methods of the Freedom quit line. Contemp Clin Trials. 2017 Aug;59:51-56. doi: 10.1016/j.cct.2017.04.011. Epub 2017 May 4. No abstract available. PMID 28479219
- [Derived] Cassidy DG, Wang XQ, Mallawaarachchi I, Wiseman KP, Ebbert JO, Blue Star JA, Aycock CA, Estevez Burns R, Jones JR, Krunnfusz AE, Halbert JP, Roy NM, Ellis JM, Williams JB, Klesges RC, Talcott GW. Tobacco quitline performance: Comparing the impacts of early cessation and proactive re-engagement on callers' smoking status at follow-up at 12 months. Tob Induc Dis. 2023 Feb 15;21:24. doi: 10.18332/tid/159125. eCollection 2023. PMID 36798676
- [Derived] Wiseman KP, Aycock CA, Mallawaarachchi I, Wang XQ, Cassidy DG, Patience MA, Little MA, Talcott GW, Klesges RC. Predictors of Re-Engagement after Relapse in a Tobacco Quit Line Intervention: Secondary Analysis from a Randomized Clinical Trial. Int J Environ Res Public Health. 2023 Jan 10;20(2):1229. doi: 10.3390/ijerph20021229. PMID 36673992